CLINICAL TRIAL: NCT05171010
Title: Geri-TBI: A Prospective Multi-center Evaluation of Geriatric Patients With Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 049.GME.2017.D
Record Dates: First submitted 2020-09-22; First posted 2021-12-28 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Other: no study-based therapeutic interventions — no study-based therapeutic interventions

SUMMARY:
This multicenter prospective observational study is designed to prospectively record data on patients who are managed per institutional standard of care. The objectives of this study are to establish an aggregate database of information on baseline clinical and demographic characteristics, medication use, markers of frailty, injury characteristics, management strategies, and outcomes following TBI in geriatric patients, determine best practices for management of geriatric patients with TBI, and establish how markers of frailty correlate with outcome in geriatric patients with TBI.

DETAILED DESCRIPTION:
This is a prospective multi-center observational study of geriatric patients with TBI. Data collected will be purely observational and involve no study-based therapeutic interventions or alterations in patient care. Due to the purpose of this study being the creation of a registry and the absence of demographic information being collected, all patients meeting the inclusion criteria will be enrolled without informed consent. We plan to complete the data collection and analysis by 12/31/2018.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40
* CT-verified TBI

Exclusion Criteria:

1. Any other body region injury AIS >2
2. Presentation at enrolling center >24 hours after injury
3. Pregnant women
4. Prisoners

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Geriatric patients with TBI
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
CT scan | "through study completion, an average of 1 year".
  CT scan-verified traumatic brain injury in patients aged greater than or equal to 40

SECONDARY OUTCOMES:
Comorbidities | "through study completion, an average of 1 year".
  history of any systemic diseases like diabetes, hypertension, blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Michael Truitt, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided